CLINICAL TRIAL: NCT05665959
Title: The Effect of Reiki Therapy on Pain, Functional Status and Holistic Well-being in Patients With Knee Osteoarthritis: A Randomized Controlled Study
Brief Title: Reiki Effects on Pain, Functional Status and Holistic Well-Being in Patients With Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Other Study IDs: 129
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis; Pain
Keywords: Reiki; functional status; pain; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reiki Group: Patient Information Form (PIF), Visual Analog Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Holistic Well-Being Scale (HWS) were administered to the Reiki group. After the pretests of the patients were completed, the primary investigator with Reiki second degree applied Reiki therapy to the patients for 40 minutes. On the second and third days, she applied distant reiki. After 3 days and 10 days after the patients were included in the study, the post-tests were performed by calling the patients.
  Interventions: Other: Reiki
- Control Group: Patient Information Form (PIF), Visual Analog Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Holistic Well-Being Scale (HWS) were administered to the control group. After 3 days and 10 days after the patients were included in the study, the post-tests were performed by calling the patients.

INTERVENTIONS:
Other: Reiki — Reiki is based on the belief that disease occurs when an energy center is blocked, and that the energy is transmitted through touch. In distant Reiki, Reiki practitioners followed the traditional Usui Reiki protocol for distant healing.
  Groups: Reiki Group

SUMMARY:
This study aimed to examine the effect of Reiki therapy on pain, functional status and holistic well-being in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is a chronic degenerative joint disease that causes pain in individuals and negatively affects their functional status and overall well-being. Patients often benefit from non-pharmacological methods in pain control. Reiki, expressed as "universal life energy", is a kind of energy therapy that creates the appropriate conditions required by the body's natural healing system in rebalancing and recharging human energy fields. Although Reiki studies in the field of orthopedics are limited, it is revealed that Reiki improves physical function, reduces fatigue and increases emotional well-being in rheumatoid arthritis patients. Studies evaluating the effectiveness of Reiki in patients undergoing total knee replacement have evaluated that Reiki is effective in controlling postoperative pain, reducing blood pressure, respiratory rate, and state anxiety.

The study was conducted with patients with knee osteoarthritis who applied to the orthopedic outpatient clinic of a training and research hospital between June 24, 2022 and December 31, 2022. The data of the study was collected using "Patient Information Form (PIF)", "Visual Analog Scale (VAS)", "Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)" and "Holistic Well-Being Scale (HWS).

PIF, VAS, WOMAC and HWS were applied to the patients who met the inclusion criteria and agreed to participate in the study. Patients were randomized 1:1 into groups by a single therapist according to the block randomization method. There were two arms in the study; Reiki treatment (n=21) and control group (n=21). A second-degree Reiki practitioner applied Reiki to the patients for 40 minutes. On the second day and the third day, 30 minutes distant Reiki were applied to the patients. In the control group, nothing was done. Post-tests were applied to all patients 3 days and 10 days after they were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2-3 osteoarthritis according to the Kellgren Lawrence scale,
* Patients aged 40 and over

Exclusion Criteria:

* Those who have difficulty in responding to the data collection form to be used in the research and have problems in understanding and communicating Turkish,
* Those who refuse to answer the Reiki application and data collection tools,
* Those who want to leave at any stage of the research or cannot be reached by phone,
* Those who underwent an application such as physical therapy, intraarticular injection or prolotherapy during the research process,
* Those who used any Complementary and Alternative Method (CAM) in the last 6 months were excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included who has grade 2 or three knee osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | Baseline
  The form created by the researchers included 11 questions covering the sociodemographic characteristics of the patients such as gender, age, marital status and the characteristics of the disease/treatment process.
Visual Analog Scale | Change from baseline Visual Analog Scale at 3 days and 10 days
  It is a reliable and easily applicable scale used to measure the severity of pain in patients, accepted in the world literature. The scale, which was used to digitize the values that could not be measured numerically, was used to evaluate the pain intensity of the patients. A minimum of 0 and a maximum of 10 points can be obtained from the scale. In addition, high scores indicate increased pain intensity.
Western Ontario and McMaster Universities Osteoarthritis Index | Change from baseline Western Ontario and McMaster Universities Osteoarthritis Index at 3 days and 10 days
  It is a valid and reliable index that is widely used for the evaluation of patients with osteoarthritis. The WOMAC Osteoarthritis index, which was validated and reliable in Turkish by Tüzün et al. in our country, consists of three sections and 24 questions in which pain, stiffness and physical function are questioned. Each question was scored on a Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The maximum scores that can be obtained from the index are 20 for the pain subgroup, 8 for stiffness, and 68 for physical function. High scores indicate increased pain and stiffness and impaired physical function.
Holistic Well-Being Scale | Change from baseline Holistic Well-Being Scale at 3 days and 10 days
  The scale is graded from disagree (1) to completely agree (10). The minimum score of the scale is 10 and the maximum score is 260, and as the score obtained from the scale increases, holistic well-being improves.

CONTACTS AND LOCATIONS:
Overall Officials: Nursemin Unal, Principal Investigator — Ankara Medipol University
Locations (1):
- Nursemin Ünal, Ankara, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Notte BB, Fazzini C, Mooney RA. Reiki's effect on patients with total knee arthroplasty: A pilot study. Nursing. 2016 Feb;46(2):17-23. doi: 10.1097/01.NURSE.0000476246.16717.65. PMID 26760383
- [Background] Topdemir EA, Saritas S. The effect of Acupressure and Reiki application on Patient's pain and comfort level after laparoscopic cholecystectomy: A randomized controlled trial. Complement Ther Clin Pract. 2021 May;43:101385. doi: 10.1016/j.ctcp.2021.101385. Epub 2021 Apr 2. PMID 33836405
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997